CLINICAL TRIAL: NCT06384872
Title: Effect of Foam Properties and Cushioning Position of Running Shoes on Injury Risk in Leisure-time Runners: A Randomized Trial
Brief Title: Effect of Shoe Cushioning Position and Properties on Running-related Injury Risk
Acronym: RRI_Interv5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: DECATHLON SA (Unknown)
Responsible Party: Principal Investigator, Laurent Malisoux, PhD, Group leader, Luxembourg Institute of Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 230042_RRI_Interv5
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Running-related Injury
Keywords: Bodymass; Musculoskeletal; Prevention; Epidemiology; Footwear; Cushioning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be stratified according to their sex. Two pre-established randomization list will be prepared by a statistician not involved in any other part of the study before the beginning of the study. To ensure allocation concealment, the study groups as well as the shoes will be coded and the randomization lists will be uploaded in the electronic system by an IT specialist who will not be involved in any other part of the study. The electronic system will provide the investigator with a study group code for each participant, according to the randomization lists. The investigator will upload the shoe ID according to shoe size and study group so that a cross validation will be performed by the electronic system. The investigators in charge of the recruitment, follow-up and data validity check, as well as the participants, will be blinded regarding the shoe version distributed. The shoe code will be broken after completion of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hard-Hard cushioned running shoes (Experimental): Running shoes with cushioned properties (linear equivalent stiffness) as follow: about 60 and 80 N/mm at the rear and forepart of the shoe, respectively.
  Interventions: Other: Shoe Cushioning Position and Properties
- Soft-Hard cushioned running shoes (Experimental): Running shoes with cushioned properties (linear equivalent stiffness) as follow: about 40 and 80 N/mm at the rear and forepart of the shoe, respectively.
  Interventions: Other: Shoe Cushioning Position and Properties
- Soft-Soft cushioned running shoes (Experimental): Running shoes with cushioned properties (linear equivalent stiffness) as follow: about 40 and 50 N/mm at the rear and forepart of the shoe, respectively.
  Interventions: Other: Shoe Cushioning Position and Properties

INTERVENTIONS:
Other: Shoe Cushioning Position and Properties — The three running shoe models will be exactly the same, except for their foam properties at the rear and forepart of the shoe, which will differ by 33 and 37%, respectively, while remaining within the range of values of shoes available on the market (linear equivalent stiffness: about 40 to 60 and 50 to 80 N/mm, at the rear and forepart of the shoe, respectively). We expect a difference in shoe weight lower than 30 g between the three versions (for size 42). The difference in cushioning properties between shoe versions will be created by modifying the type of foam and the foaming process.

SUMMARY:
The main purpose of this project is to investigate the influence of cushioning material at both the rear and the forepart of running shoes on musculoskeletal complaints in leisure-time runners. Therefore, the objectives are to investigate if

1. "Extra soft" cushioning materials can reduce injury risk compared to stiffer materials;
2. Cushioning under the forepart of the shoe also influences injury risk, independently of the cushioning at the rear part;
3. Effects of cushioning material and position depend on the runner's body mass;
4. Perception of cushioning is related to both shoe cushioning and injury risk;
5. Other weight-bearing locomotion activities (i.e., number of steps per day besides running practice) represents an independent risk factor for running-related injury.

This study consists in a 6-month intervention trial during which leisure-time runners are required to follow their usual training schedule. Before the beginning of the study, the participants will receive a pair of running shoes. The three running shoe models will be exactly the same, except for their foam properties at the rear and forepart of the shoe, which will differ by 33 and 37%, respectively. The study shoes will be administered through random allocation. The participants will be required to use these shoes for all running sessions, and only for running activities.

Participants will first fill out a baseline questionnaire. During the intervention, data on running practice will be downloaded from sports watches via their respective app. Information on the use of the study shoes will be collected via a weekly questionnaire. Participants will be asked to fill out a weekly questionnaire on any musculoskeletal complaints experienced during the past 7 days. A questionnaire on the perception of cushioning will be filled in by the participants at three time points (after 5h of running, 25h of running, and at the end of follow-up).

Primary hypothesis:

- Greater shock absorption properties at the rear part of running shoes are associated with a lower injury risk in recreational runners.

Secondary hypothesis:

* Greater shock absorption properties under the forepart of the shoe are also associated with lower injury risk in recreational runners.
* Runners with low body mass experience a lower injury risk in shoes with greater shock absorption properties.
* Greater perceived cushioning is related to lower injury risk.

DETAILED DESCRIPTION:
Study design:

The design of this study is a randomized trial with an intervention period of six months. Running footwear is provided by a renowned sport equipment manufacturer working in close collaboration with the Physical Activity, Sport and Health (PASH) research group of the Luxembourg Institute of Health (LIH). PASH will be responsible for the management and execution of the study, including random allocation of the study shoes, recruitment and follow-up of the participants, as well as data management and analysis. The study design is based on the comparison of three running shoe versions, which differ with respect to their foam properties and cushioning position (i.e., rear and forepart of the shoe). The cushioning properties at the rear and forepart of the three shoe versions will be within the range of values of models available on the market.

Participants:

Healthy leisure-time runners will be recruited through advertising in local newspapers and press releases within Luxembourg, as well as via social media during the months of March 2025 to August 2025. The benefits for the participants are highlighted during the recruitment phase, and are as follows: 1) a free pair of running shoes, and 2) a brief report on the main findings of the study. However, participants will be made aware that they will randomly receive one of the three study shoe versions to be worn during the intervention period for all their running activities.

Volunteers willing to take part in the study will be invited to follow the process described hereafter:

* Volunteers have to register on the electronic system that will be specifically designed for the study, and specify that they wish to enroll for the present study. The inclusion/exclusion criteria and study requirements will be reminded at this stage of the registration process.
* Volunteers will receive the full information of the study, and informed consent containing the full name of the participants.
* Volunteers must declare that they freely consent to participate in the study by checking the appropriate boxes.
* Volunteers will have to fill in a baseline questionnaire.
* Volunteers will have to set an appointment with the research team via the electronic system.

Sample size:

A sample size calculation for Cox regression was used to determine the number of participants needed for the primary hypothesis of the study. With an alpha of 0.05 and a power of 80%, an average injury rate of 30% (see definition of the main outcome below), an expected HR=1.50 between groups, 33% of participants randomized to each shoe group and an expected drop-out rate of 10%, the total number of participants required is 1068.

Intervention:

The study shoes are prototypes derived from a model available on the market (Kiprun KS 500.2) and will be anonymized for the purpose of this trial. The sole of the shoes will be customized for the purpose of the study. The three running shoe models will be exactly the same, except for their foam properties at the rear and forepart of the shoe, which will differ by 33 and 37%, respectively, while remaining within the range of the shoes available on the market (linear equivalent stiffness: 40 to 60 and 50 to 80 N/mm, at the rear and forepart of the shoe, respectively). We expect a difference in shoe weight lower than 30 g between the three versions (for size 42). The difference in cushioning properties between shoe versions will be created by modifying the type of foam and the foaming process. A set of shoes will be tested for cushioning properties by the manufacturer to provide accurate data on the technical specifications (stiffness and dissipated energy).

* Model 1: "Hard" - about 60 and 80 N/mm at the rear and forepart of the shoe, respectively.
* Model 2: "Mixed" - about 40 and 80 N/mm at the rear and forepart of the shoe, respectively.
* Model 3: "Soft" - about 40 and 50 N/mm at the rear and forepart of the shoe, respectively.

The main hypothesis will be tested comparing the Mixed shoe version with the Hard shoe version, while the secondary hypothesis will be tested comparing the Soft shoe version with both the Hard and Mixed shoe versions.

Stratified randomization:

Participants will be randomized at a 1:1:1 ratio to one of the three treatment arms. A block randomization (block size 12) will be performed. Randomization will be stratified by sex, as the latter influences body mass. Based on data from previous studies, it is expected that the study population will include about 40% of women. Two pre-established randomization lists will be provided by a statistician (LIH) not involved in any other part of the study before the beginning of recruitment. The participant identification number will be composed of 4 digits: first digit corresponding to the participant's sex (1=female, 2=male) followed by 3 digits corresponding to the randomization number.

Data collection:

Participants will have to fill in a baseline questionnaire that aims to collect information regarding demographics, running experience, training habits, running competitions performed and injury history. The recruitment phase of this project will last from March 2025 until August 2025. The follow-up period will start as soon as the participants have received their study shoes and will last for 6 months. This means that the data collection phase will finish at the latest on the 28th of February 2026.

Once a participant receives his/her pair of study shoes, the intervention period begins for that participant. During this intervention period, the participants are required to use the study shoes for all their running activities, to continue their usual or follow their planned training schedule, and to fill out the weekly questionnaire on musculoskeletal complaints, as well as on the use of the study shoes during the follow-up.

Data on running practice will be downloaded from sports watches (i.e., Garmin, Polar and Suunto) via their respective applications. Data can also be downloaded from other applications (GPX files from any activity tracker with GPS) and subsequently uploaded into the electronic system "STRIDE". Information on the use of the study shoes will be collected via a weekly questionnaire.

Study participation will be terminated and the participant will be right-censored if he/she does not fill in the weekly injury form for 2 consecutive weeks, does not reply (or react) to the automatic reminders (2 days after the initial invitation), and could not be reached by phone by the research team (2 attempts). Indeed, a critical aspect for the validity of the study is to verify that the injury (the main outcome) is not the reason for dropping out. Therefore, we will contact these participants to confirm that they reported all injury before termination of the investigation.

Participants will be asked to fill out a weekly questionnaire on any physical complaints experienced during the past 7 days (the Oslo Sports Trauma Research Centre (OSTRC) Overuse Injury Questionnaire). On top of the four basic questions, information regarding the following is required: data of first onset, sports discipline, anatomical location, type of injury, new / recurrent / subsequent event, and estimated return date to full participation. Individual e-mail reminders will be sent to the participants who do not fill out a weekly questionnaire. Personal phone calls will be made if the participants do not react to the e-mail reminders and if the reported information in the injury form is found to be inconsistent.

Study outcomes:

Primary outcome

- First running-related injury occurring during the follow-up, and defined as any running-related physical complaint in the lower limbs or lower back region that causes a restriction on or stoppage of running (distance, speed, duration, or training) for at least seven days. Practically, this corresponds to injury forms where the participant answered option 3 or 4 in question 1, or option 1, 2 or 3 in question 2 or question 3 of the OSTRC-O questionnaire.

Secondary outcomes:

* First one-day time loss running-related injury: Any running-related physical complaint in the lower limbs or lower back region that causes a restriction on or stoppage of running (distance, speed, duration, or training) for at least one day. More specifically, this correspond to injury forms with option 3 or 4 in question 1, or option 1, 2 or 3 in question 2 or question 3 of the OSTRC-O questionnaire, without any minimal duration.
* First running-related musculoskeletal complaint: Any physical complaint including pain, ache, joint instability, stiffness, or any other complaint resulting from participating in running activities, including but irrespective of the need of medical attention (seeking care from medical practitioner) or time-loss (inability to complete a running training session or participate in one or more days after the onset of injury). More specifically, injury forms with option 2 in question 1 of the OSTRC questionnaire will also be considered as outcome of interest in this case;
* First substantial running-related injury: Injury forms where the participant answered options 3 or 4 in question 2 or question 3 of the OSTRC-O questionnaire.
* First overuse running-related injury: Injury forms where the participant reported complaints with obvious acute mechanism such as ankle sprain will be excluded (considered as competing risk).

Statistical analysis:

Descriptive data for the personal and training-related characteristics will be presented as count and percentage for dichotomous variables, and as mean and standard deviation, or as median and range, for normally and non-normally distributed continuous variables, respectively. Average sport-related characteristics will be computed for each participant over their specific period of observation. Shock absorption properties of the three shoes versions (measured and provided by Decathlon) will be compared using an Analysis of Variance.

We will calculate the injury incidence as number of injuries per 1000 hours of running exposure for each outcome. We will calculate the injury prevalence each week by dividing the number of participants that reported an injury by the number of respondents that week for each outcome. We will then calculate the average weekly prevalence for each outcome and separately for the main anatomic locations.

Competing-risks regression models will be used to investigate the effect of shoe version, body mass and other possible risk factors by estimating the subdistribution hazard, according to Fine and Gray. Date of inclusion and date of injury or censoring will be basic data used to calculate the time at risk, which is expressed in hours spent running and defined as the time-scale. Participants will be right-censored if lost to follow-up or at the end of the intervention period. Average sport-related characteristics will be computed for each participant over their specific period of observation. The assumption of proportional hazards was evaluated using log-minus-log plots and Schoenfeld's global test. First, unadjusted subdistribution hazards will be estimated for shoe versions, body mass and other potential risk factors such as training-related characteristics. Subsequently, the variables with a P value <0.200, as well as well-established potential confounders, will be included in the adjusted model to determine whether shoe cushioning is associated with injury risk. The recommendation for using at least ten injuries per predictor variable included in the regression analysis will be strictly followed. Finally, a stratified analysis will be performed to investigate if the effect of shoe cushioning on injury risk is modified by body mass. Participants will be classified as light or heavy runners using the median value of body mass as cut-off, independently in men and women. SHRs and their 95% confidence intervals (CI) will be first determined for each stratum (with the reference being the stratum with the lower risk). Then, SHRs and their 95% CI will be computed within strata to determine both the effect of shoe version within each body mass category, and the effect of body mass within each shoe group.

Sensitivity analysis First, we will exclude the participants who sustained an injury over the first two weeks to investigate the potential impact of the transition to the study shoe on the findings. Second, depending on the compliance of the participants to the intervention (i.e., use of the study shoes for each running session), we will exclude the participants who did not use the study shoes for (e.g.) minimum 50% of their running sessions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Willing to use the study shoes for each running training session, and only for running activities
* Use a sports watch for training data recording
* Accept to give access to running data via a Garmin Connect, Polar Flow or Suunto account, or accept to upload the GPX file (downloaded from another system) into the electronic system "STRIDE" for every running session
* Signed electronic Informed Consent provided

Exclusion Criteria:

* Women who are pregnant
* Any contraindication to running training including cardiovascular/respiratory disease or running impeding injury/condition at the time of initial inclusion;
* A history of surgery to the lower limbs or the lower back within the previous 12 months or any degenerative conditions;
* The use of orthopedic insoles for physical activity;
* Any running injury (a physical pain or complaint related to running practice that causes the runner to interrupt or modify his/her training for at least one week) over the last month.

No limitation will be set regarding running experience, running level (performance), body mass or body mass index.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1068 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
First running-related injury with a duration of minimum one week | 6 months
  First running-related injury occurring during the follow-up, and defined as any running-related physical complaint in the lower limbs or lower back region that causes a restriction on or stoppage of running (distance, speed, duration, or training) for at least seven days. Practically, this corresponds to injury forms where the participant answered option 3 or 4 in question 1, or option 1, 2 or 3 in question 2 or question 3 of the OSTRC-O questionnaire, with a duration of minimum one week.

SECONDARY OUTCOMES:
First one-day time loss running-related injury | 6 months
  Any running-related physical complaint in the lower limbs or lower back region that causes a restriction on or stoppage of running (distance, speed, duration, or training) for at least one day. More specifically, this correspond to injury forms with option 3 or 4 in question 1, or option 1, 2 or 3 in question 2 or question 3 of the OSTRC-O questionnaire, without any minimal duration.
First running-related musculoskeletal complaint to the lower limb | 6 months
  Any musculoskeletal complaint including pain, ache, joint instability, stiffness, or any other complaint resulting from participating in running activities, including but irrespective of the need of medical attention (seeking care from medical practitioner) or time-loss (inability to complete a running training session or participate in one or more days after the onset of injury). More specifically, injury forms with option 2 in question 1 of the OSTRC questionnaire will also be considered as outcome of interest in this case.
First substantial running-related injury | 6 months
  Injury forms where the participant answered options 3 or 4 in question 2 or question 3 of the OSTRC-O questionnaire.
First overuse running-related injury | 6 months
  Injury forms where the participant reported complaints with obvious acute mechanism such as ankle sprain will be excluded (considered as competing risk).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Malisoux, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute of Health, Strassen, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarsen B, Bahr R, Myklebust G, Andersson SH, Docking SI, Drew M, Finch CF, Fortington LV, Haroy J, Khan KM, Moreau B, Moore IS, Moller M, Nabhan D, Nielsen RO, Pasanen K, Schwellnus M, Soligard T, Verhagen E. Improved reporting of overuse injuries and health problems in sport: an update of the Oslo Sport Trauma Research Center questionnaires. Br J Sports Med. 2020 Apr;54(7):390-396. doi: 10.1136/bjsports-2019-101337. Epub 2020 Feb 14. PMID 32060142
- [Background] Malisoux L, Delattre N, Urhausen A, Theisen D. Shoe Cushioning Influences the Running Injury Risk According to Body Mass: A Randomized Controlled Trial Involving 848 Recreational Runners. Am J Sports Med. 2020 Feb;48(2):473-480. doi: 10.1177/0363546519892578. Epub 2019 Dec 26. PMID 31877062
- [Derived] Malisoux L, Urhausen A, Flores N, Theisen D, Morio C. Running shoe cushioning properties at the rearfoot and forefoot and their relationship to injury: study protocol for a randomised controlled trial on leisure-time runners. BMJ Open Sport Exerc Med. 2024 Oct 11;10(4):e002217. doi: 10.1136/bmjsem-2024-002217. eCollection 2024. PMID 39415882
- See also: Research group webpage — https://www.lih.lu/en/research-scope/research-department/department-of-precision-health/physical-activity-sport-and-health/
- See also: Project page — https://stride.lih.lu